CLINICAL TRIAL: NCT06135181
Title: Randomized, Single-blind, Placebo-controlled, Escalating Single-dose Study of Safety, Tolerability, and Pharmacokinetics of Intravenously Administered BAY 1747846 in Healthy Chinese Men
Brief Title: A Study to Learn More About the Safety and the Blood Level of BAY1747846 Given as Injection Into the Vein at Increasing Single Doses in Chinese Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 19730
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Contrast Enhancement in Magnetic Resonance Imaging; Healthy Volunteers
Keywords: Safety; Pharmacokinetics

STUDY DESIGN:
Intervention Model Description: Parallel-group, consecutive cohort, escalating single-dose study design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.03 mmol Gd/kg BAY1747846 and matching placebo (Experimental): 12 healthy male participants were planned to be enrolled into this arm, 9 on BAY1747846 and 3 on placebo
  Interventions: Drug: Gadoquatrane (BAY1747846) 0.03 mmol Gd/kg; Drug: Matching placebo
- 0.1 mmol Gd/kg BAY1747846 and matching placebo (Experimental): 12 healthy male participants were planned to be enrolled into this arm, 9 on BAY1747846 and 3 on placebo
  Interventions: Drug: Gadoquatrane (BAY1747846) 0.1 mmol Gd/kg; Drug: Matching placebo

INTERVENTIONS:
Drug: Gadoquatrane (BAY1747846) 0.03 mmol Gd/kg — 0.03 mmol Gd/kg by intravenous injection (at 2 mL/s)
  Arms: 0.03 mmol Gd/kg BAY1747846 and matching placebo
Drug: Gadoquatrane (BAY1747846) 0.1 mmol Gd/kg — 0.1 mmol Gd/kg by intravenous injection (at 2 mL/s)
  Arms: 0.1 mmol Gd/kg BAY1747846 and matching placebo
Drug: Matching placebo — 0.9% sodium chloride by intravenous injection (at 2 mL/s)

SUMMARY:
The goal of this clinical study was to learn more about BAY1747846 compared to placebo when given as an injection into the vein in Chinese healthy male participants:

* the safety of BAY1747846 when given at increasing single doses
* the level of BAY1747846 in the blood over time when given at increasing single doses.

To answer the first question, the researchers compared the number and severity of medical problems the Chinese participants had after receiving BAY1747846 at increasing doses and placebo respectively. Doctors kept tracking of all medical problems that happened in the study, even if they did not think they might be related to the study treatments.

To answer the second question, the researchers determined:

* the (average) total level of BAY1747846 in the blood, also called AUC
* the (average) highest level of BAY1747846 in the blood, also called Cmax
* how BAY1747846 is removed from the blood, also called clearance (CL).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study specific tests or procedures
* Chinese male between 18 and 45 years (inclusive) at screening visit
* Body mass index (BMI): 18.5 to 30.0 kg/m² (inclusive)
* Body weight (bw): 50 to 90 kg (inclusive)
* Participants of reproductive potential must agree to use adequate contraception whenever having sexual intercourse with a woman of child-bearing potential. This applies for the time period from signing of the ICF to at least 1 week after treatment. The definition of adequate contraception will be based on the judgment of the investigator and on local requirements
* Healthy, based on medical history, physical examination, electrocardiography (ECG), and laboratory tests

Exclusion Criteria:

* Use of systemic or topically active medication or herbal remedies, prescription or non-prescription, from screening to the first drug administration (only use of contraceptives and occasional use of paracetamol, aspirin or ibuprofen is permissible)
* Any severe disease within the last 4 weeks prior to the first study drug administration
* Any clinically relevant finding at the physical examination and chest X ray (posterior-anterior) examination
* Any clinically relevant deviation from reference ranges of the laboratory parameters at screening or alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin exceeding the upper limit of normal range (ULN) by more than 10%, or creatinine above the ULN, or hemoglobin below 12 g/dL
* Vital signs: Pulse rate <50 or >90beats/min, Systolic blood pressure <100 or ≥140 mmHg, Diastolic blood pressure <60 or ≥90 mmHg, or other abnormal vital signs
* Any known disposition for allergic, anaphylactoid, hypersensitivity or idiosyncratic reactions, e.g. any history of clinical signs of hypersensitivity reaction to any agent (including, but not limited to, any allergen, food, drug, chemical, or contrast agent)
* Family history of hypersensitivity reaction to contrast agent
* Regular alcohol consumption equivalent to >20 g alcohol per day within 3 months prior to screening
* Smokers who smoke more than 5 cigarettes per day within 3 months prior to screening and/or who cannot refrain from smoking from screening until the end of hospitalization
* Criteria which in the opinion of the investigator preclude participation for scientific reasons, for reasons of compliance, or for reasons of the participant's safety

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAE) | From drug administration up to 7 days after end of test drug administration (from day 1 to day 8)
  Including severity of TEAE

SECONDARY OUTCOMES:
Cmax | Pre-dose, on Day 1, Day 2, Day 3 and Day 4
  Cmax: Maximum observed drug concentration in measured matrix after single dose administration
AUC | Pre-dose, on Day 1, Day 2, Day 3 and Day 4
  AUC: Area under the concentration vs. time curve from zero to infinity after single dose in case AUC cannot be determined reliably for all participants, AUC will be replaced by AUC(0-tlast)
CL | Pre-dose, on Day 1, Day 2, Day 3 and Day 4
  CL: Total body clearance of drug
CL/bw | Pre-dose, on Day 1, Day 2, Day 3 and Day 4.
  CL/bw: Total body clearance of drug normalized by body weight

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/19730